CLINICAL TRIAL: NCT07082166
Title: Comparison of the Effects of Connective Tissue Massage and Extracorporeal Shock Wave Therapy (ESWT) in Patients With Fibromyalgia Syndrome
Brief Title: Comparison of the Effects of Fibromyalgia Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ilknur Mazı, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: ISTANBUL-UC-MAZI
Record Dates: First submitted 2025-07-13; First posted 2025-07-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
Keywords: FIBROMYALGIA SYNDROME; Connective Tissue Massage; Extracorporeal Shock Wave Therapy; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTM GROUP: ESWT GROUP

SUMMARY:
Massage therapy, one of the complementary and alternative treatments, is commonly used for fibromyalgia syndrome (FMS). It may help improve pain, anxiety, depression, and sleep disorders through the complex interaction of physical and mental mechanisms. Although studies have investigated massage and extracorporeal shock wave therapy (ESWT) separately, there is currently no study directly comparing these two treatment methods.

In this study, we plan to use massage therapy to reduce pain, stiffness, fatigue, and sleep difficulties in individuals with FMS. The aim is to evaluate the effects of both connective tissue massage and ESWT on fibromyalgia symptoms, with a focus on pain, fatigue, sleep disturbances, health status, and quality of life.

We also aim to compare the effectiveness of these two non-pharmacological interventions in enhancing general well-being and encouraging participation in daily life. Additionally, we hope this research will contribute to clinical practice by evaluating the potential benefits of connective tissue massage, a safe and cost-effective method.

DETAILED DESCRIPTION:
General Information

Fibromyalgia syndrome (FMS) is one of the most common conditions affecting muscles and is characterized by pain, stiffness, and tenderness in muscles, tendons, and joints. Despite years of research, no definitive cause or pathophysiology of FMS has been identified. It is believed that genetic and environmental factors, as well as both peripheral and central mechanisms, may play a role in the development of widespread pain and pain sensitivity in individuals with fibromyalgia. FMS is often associated with symptoms such as decreased physical capacity, fatigue, sleep disorders, gastrointestinal issues, and psychiatric conditions including depression. Pain and other symptoms interfere with daily functioning, work, and social activities, resulting in reduced quality of life.

Various treatment approaches are available for patients with FMS. Both pharmacological and non-pharmacological methods are used in its management. Treatment options include medications such as tricyclic antidepressants, exercise, acupuncture, manual/manipulative therapies, and mind-body approaches. Studies on exercise suggest that moderate-to-high intensity physical activity may be effective. Antidepressants have been found helpful in increasing serotonin levels and thereby alleviating fibromyalgia symptoms. Chiropractic care and acupuncture have also been explored as potential management strategies.

Connective Tissue Massage (CTM) Massage therapy is widely used as a complementary and alternative treatment in fibromyalgia. Through the complex interaction of physical and psychological mechanisms, it may improve pain, anxiety, depression, and sleep disturbances. When applied to soft tissues and connective tissue, massage may induce local biochemical changes that contribute to improved muscle flexibility and modulation of local blood and lymphatic circulation.

Connective tissue massage, one of the manual therapy techniques used for FMS, involves short and long tractions on the connective tissue that may mechanically stimulate mast cells. This may help reduce sympathetic activity and promote vasodilation. As a result, parasympathetic activity increases and supports improved circulation.

Extracorporeal Shock Wave Therapy (ESWT) Extracorporeal shock wave therapy is a non-invasive physical method developed from extracorporeal shock wave lithotripsy. While initial studies focused on kidney stones, recent research on the musculoskeletal system has shown that shock waves may positively affect various tissues, including bones and soft tissues.

Materials and Methods

Participants Patients diagnosed with FMS by a rheumatologist according to ACR criteria and referred to the Department of Physiotherapy and Rehabilitation will be assessed for eligibility.

Assessment Tools Demographic and clinical information will be collected using a custom-designed form developed by the researchers. This form includes gender, age, height, weight, education level, and medical history (e.g., chronic diseases, past injuries, eating disorders). Participants will be instructed on how to complete the form, and data will be used for scientific purposes only.

Evaluation Methods

Pain will be assessed using the McGill Pain Questionnaire, which includes a scale from "no pain" to "unbearable pain" and body diagrams for pain localization.

Quality of life will be evaluated with the Nottingham Health Profile, measuring the impact of health on function and well-being.

Fibromyalgia Impact will be measured by the Fibromyalgia Impact Questionnaire, assessing physical health, work status, depression, anxiety, sleep, pain, fatigue, stiffness, and well-being. Higher scores indicate lower functioning.

Sleep quality will be assessed with the Pittsburgh Sleep Quality Index, including components such as sleep duration, latency, medication use, and daytime functioning.

Mechanical pain sensitivity will be measured using an algometer. Pressure will be applied to tender points until the participant indicates pain. The procedure will be repeated for reliability, and pressure will be recorded in Newton/cm².

Anxiety will be evaluated using the State-Trait Anxiety Inventory, where higher scores indicate greater anxiety.

Interventions and Statistical Methods Participants will be randomly assigned to two groups. Both groups will receive treatment on the same anatomical regions. One group will receive connective tissue massage, and the other will receive extracorporeal shock wave therapy. Both groups will also engage in a walking program and posture exercises. Evaluations will be conducted at baseline, post-treatment, and at follow-up.

Treatment Protocols

Connective Tissue Massage: Administered with the patient in a prone position. Areas treated include the lumbosacral, lower thoracic, scapular, interscapular, and cervical regions. The therapist will use finger traction techniques. Sessions will last approximately 30 minutes.

Extracorporeal Shock Wave Therapy: Applied with the patient in the same position using a medical device. Parameters include defined pressure levels and a specific number of pulses per session. Sessions will be brief.

Statistical Analysis Data will be analyzed using SPSS software. Normality will be tested, and appropriate parametric or non-parametric tests will be used. Variables will be presented as means, standard deviations, confidence intervals, and percentages. Between-group differences will be analyzed with t-tests and chi-square tests. Pre- and post-treatment changes will be evaluated with paired tests. Statistical significance will be set at p < 0.05. Effect sizes will be calculated and categorized as small, medium, or large.

Power Analysis Sample size was calculated using power analysis software. Based on expected effect sizes and desired power, the required number of participants per group was determined. The final sample size was increased to account for potential dropouts.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia syndrome
* Aged between 18 and 60 years
* Female gender
* Symptoms present for at least 6 months
* Willing to participate in the study
* Literate

Exclusion Criteria:

* History of rheumatologic, neurologic, psychiatric, or systemic disease
* Pregnancy or lactation
* Prior treatment with massage or ESWT
* History of acute infection, trauma, or surgery
* History of cancer
* Use of painkillers or antidepressants
* Any medical condition that prevents participation in physical activity

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients residing in Istanbul who applied to our center, both employed and unemployed, were included
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
3.1. Pain (Mcgill) | 6 WEEK
  Higher scores indicate more severe pain. Description: Consists of 15 pain descriptors (11 sensory, 4 affective), each rated on a scale from 0 (none) to 3 (severe), plus a Visual Analog Scale (VAS) and Present Pain Intensity (PPI)

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 6 week
  Higher scores indicate greater disease impact and worse functional status. Description: Measures physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gerontechnology Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No